CLINICAL TRIAL: NCT01342965
Title: A Multicenter, Open-label, Randomized Phase III Study to Evaluate the Efficacy and Safety of Erlotinib (Tarceva®) Versus Gemcitabine/Cisplatin as the First-line Treatment for Stage IIIB/IV Non-small Cell Lung Cancer (NSCLC) Patients With Mutations in the Tyrosine Kinase Domain of Epidermal Growth Factor Receptor (EGFR) in Their Tumors
Brief Title: A Study of Erlotinib (Tarceva) Versus Gemcitabine/Cisplatin as First-line Treatment in Patients With Non-small Cell Lung Cancer With EGFR Mutations
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YO25121
Record Dates: First submitted 2011-04-26; First posted 2011-04-27 (Estimated); Results first posted 2015-02-24 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2015-02

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Drug Therapy

ARMS (2):
- Erlotinib (Experimental): Participants received erlotinib 150 mg orally once daily until progressive disease or unacceptable toxicity.
  Interventions: Drug: Erlotinib
- Chemotherapy (Active Comparator): Participants received gemcitabine 1250 mg/m^2 intravenously (IV) on Days 1 and 8 and cisplatin 75 mg/m^2 IV on Day 1 of every 3 week cycle until disease progression, unacceptable toxicity, or a total of 4 cycles, whichever came first.
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Erlotinib — Erlotinib was supplied as tablets.
  Other Names: Tarceva
  Arms: Erlotinib
Drug: Chemotherapy — Cisplatin and gemcitabine were locally sourced with commercial products.
  Arms: Chemotherapy

SUMMARY:
This open-label, randomized, parallel arm study assessed the efficacy and safety of Tarceva (erlotinib) versus gemcitabine/cisplatin combination chemotherapy as first-line treatment in patients with stage IIIB/IV non-small cell lung cancer with epidermal growth factor receptor (EGFR) mutations in their tumours. Patients were randomized to receive either Tarceva 150 mg orally daily or 3-week cycles of gemcitabine 1250 mg/m^2 intravenously (iv) on Days 1 and 8 plus cisplatin 75 mg/m^2 iv on Day 1.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants, ≥ 18 years of age.
* Locally advanced or recurrent (stage IIIB) or metastatic (stage IV) non-small cell lung cancer.
* Presence of epidermal growth factor receptor (EGFR) mutations in tumours.
* Measurable disease according to Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1 criteria.
* European Cooperative Oncology Group (ECOG) performance status ≤ 2.

Exclusion Criteria:

* Prior exposure to agents directed at the human epidermal receptor (HER) axis (eg, but not limited to erlotinib, gefitinib, cetuximab, or trastuzumab).
* Prior chemotherapy or systemic anti-neoplastic therapy for advanced disease.
* Lack of physical integrity of the upper gastrointestinal tract, or malabsorption syndrome, or inability to take oral medication, or active gastroduodenal ulcer disease.
* Any inflammatory changes of the surface of the eye.
* ≥ Grade 2 peripheral neuropathy.
* History of any other malignancies within 5 years, except for adequately treated carcinoma in situ of the cervix or basal or squamous cell skin cancer.
* Brain metastasis or spinal cord compression that has not yet been definitely treated with surgery and/or radiation, or treated but without evidence of stable disease for at least 2 months.
* Human immunodeficiency virus (HIV) infection.
* Pregnant, nursing, or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2011-03; Primary Completion 2012-07 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (23):
- China (11):
  - Beijing
  - Changchun
  - Chongqing
  - Fuzhou
  - Guangzhou
  - Hangzhou
  - Nanjing
  - Shanghai
  - Shantou
  - Wuhan
  - Xi'an
- Malaysia (7):
  - Kampung Baharu Nilai
  - Kelantan
  - Kuala Lumpur
  - Kuala Pahang
  - Petaling Jaya
  - Petaling Jaya, Selangor
  - Pulau Pinang
- Philippines (5):
  - Davao City
  - Desmarinas City
  - Manila
  - Quezon City
  - San Juan City

REFERENCES:
- [Derived] Wen F, Zheng H, Zhang P, Hutton D, Li Q. OPTIMAL and ENSURE trials-based combined cost-effectiveness analysis of erlotinib versus chemotherapy for the first-line treatment of Asian patients with non-squamous non-small-cell lung cancer. BMJ Open. 2018 Apr 13;8(4):e020128. doi: 10.1136/bmjopen-2017-020128. PMID 29654023
- [Derived] Wu YL, Zhou C, Liam CK, Wu G, Liu X, Zhong Z, Lu S, Cheng Y, Han B, Chen L, Huang C, Qin S, Zhu Y, Pan H, Liang H, Li E, Jiang G, How SH, Fernando MCL, Zhang Y, Xia F, Zuo Y. First-line erlotinib versus gemcitabine/cisplatin in patients with advanced EGFR mutation-positive non-small-cell lung cancer: analyses from the phase III, randomized, open-label, ENSURE study. Ann Oncol. 2015 Sep;26(9):1883-1889. doi: 10.1093/annonc/mdv270. Epub 2015 Jun 23. PMID 26105600

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Erlotinib | Chemotherapy
Started | 110 | 107
Received Treatment | 110 | 104
Completed | 1 | 0
Not Completed | 109 | 107
Not completed — Death | 58 | 57
Not completed — Lost to Follow-up | 5 | 3
Not completed — Other Reasons- Unspecified | 44 | 38
Not completed — Withdrawal by Subject | 2 | 9

BASELINE CHARACTERISTICS:
Population: Full analysis set: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Erlotinib | Chemotherapy | Total
Number analyzed (Participants) | 110 | 107 | 217
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.7 (10.37) | 55.8 (10.41) | 56.3 (10.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 65 | 133
  Male | 42 | 42 | 84

OUTCOME MEASURES:

1. Primary Outcome: Investigator-assessed Duration of Progression-free Survival
Description: The duration of progression-free survival was defined as the time from randomization to disease progression (PD) or death from any cause, whichever occurs first. PD was defined as: (1) At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this may include the baseline sum). The sum must also demonstrate an absolute increase of at least 5 mm. (2) An unequivocal progression of existing non-target lesions. When the patient has measurable disease, the overall tumor burden must have increased sufficiently to merit discontinuation of therapy. When the patient has only non-measurable disease, the increase in overall disease burden should be comparable in magnitude to the increase that would be required to declare PD for measurable disease. (3) The appearance of new malignant lesions.
Time Frame: Baseline to the data cut-off date of 20 Jul 2012 (1 year, 4 months)
Population: Full analysis set: All randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Erlotinib | Chemotherapy
Number analyzed (Participants) | 110 | 107
Months | 11.0 [8.3 to NA] — The upper limit of the confidence interval could not be estimated due to too few events. | 5.5 [4.2 to 7.1]

2. Secondary Outcome: Percentage of Responders as Assessed by the Investigator
Description: A responder was defined as a participant with either a complete response (CR) or a partial response (PR), as determined using the Response Evaluation Criteria In Solid Tumors (RECIST) v1.1. A CR was defined as: (1) The disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have a reduction in the short axis to < 10 mm. (2) The disappearance of all non-target lesions and normalization of tumor marker levels. All lymph nodes must be non-pathological in size (< 10 mm in the short axis). A PR was defined as: (1) At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. (2) The persistence of 1 or more non-target lesion(s) and/or maintenance of tumor marker levels above normal limits.
Time Frame: Baseline to the data cut-off date of 19 Nov 2012 (1 year, 8 months)
Population: Full analysis set: All randomized participants.
Measure: Number; unit: Percentage of responders
Arm/Group | Erlotinib | Chemotherapy
Number analyzed (Participants) | 110 | 107
Percentage of responders | 68.2 | 39.3

3. Secondary Outcome: Percentage of Participants With Disease Control
Description: A participant with disease control was defined as a participant with either a complete response (CR), a partial response (PR), or stable disease (SD), as determined using RECIST v1.1. A CR was defined as the disappearance of all target lesions (TL). A PR was defined as at least a 30% decrease in the sum of the longest diameter of TLs taking as reference the Baseline sum longest diameter (SLD). SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest SLD since treatment started. For non-TLs, SD was defined as the persistence of 1 or more lesions. PD was defined as at least a 20% increase in the SLD of TLs, taking as reference the smallest SLD recorded since treatment started or the unequivocal progression of existing non-TLs. A SLD for all TLs will be calculated and reported as the Baseline SLD.
Time Frame: Baseline to the data cut-off date of 19 Nov 2012 (1 year, 8 months)
Population: Full analysis set: All randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Erlotinib | Chemotherapy
Number analyzed (Participants) | 110 | 107
Percentage of participants | 91.8 | 82.2

4. Secondary Outcome: Duration of Response
Description: Duration of response was defined as the time from the first documented complete response (CR) or partial response (PR) to the first documented disease progression (PD) or death, whichever occurs first. A CR was defined as the disappearance of all target lesions (TL). A PR was defined as at least a 30% decrease in the sum of the longest diameter (SLD) of TLs taking as reference the Baseline SLD. PD was defined as at least a 20% increase in the SLD of TLs, taking as reference the smallest SLD recorded since treatment started or the unequivocal progression of existing non-TLs.
Time Frame: Baseline to the data cut-off date of 19 Nov 2012 (1 year, 8 months)
Population: Full analysis set: All randomized participants. Only participants who had a complete response or partial response were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Erlotinib | Chemotherapy
Number analyzed (Participants) | 110 | 107
Months | 10.8 [7.0 to 12.6] | 4.2 [2.8 to 5.4]

5. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from the date of randomization to the date of death from any cause.
Time Frame: Baseline to the end of the study (3 years, 1 month)
Population: Full analysis set: All randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Erlotinib | Chemotherapy
Number analyzed (Participants) | 110 | 107
Months | 28.9 [25.8 to 30.5] | 27.1 [25.4 to 30.9]

6. Secondary Outcome: Safety: Incidence of Adverse Events
Time Frame: 36 months
Reporting Status: Not Posted

7. Secondary Outcome: Quality of Life: Functional Assessment of Chronic Illness Therapy - Lung (FACIT-L) Questionnaire
Time Frame: approximately 21 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Safety analysis set: All participants who had received at least 1 dose of study medication.
Arm/Group | Erlotinib | Chemotherapy
Serious Adverse Events (participants affected / at risk) | 22/110 | 16/104
Other Adverse Events (participants affected / at risk) | 99/110 | 96/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=110) | Chemotherapy (N=104)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 3
Gastroenteritis (Infections and infestations) | 2 | 1
Pneumonia (Infections and infestations) | 3 | 0
Abscess limb (Infections and infestations) | 1 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0
Haemorrhoid infection (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 1 | 0
Nail bed infection (Infections and infestations) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 2
Thrombosis (Vascular disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0
Blood glucose increased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Bone erosion (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Spinal cord compression (Nervous system disorders) | 1 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0
Haemorrhoid operation (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=110) | Chemotherapy (N=104)
Nausea (Gastrointestinal disorders) | 5 | 60
Vomiting (Gastrointestinal disorders) | 7 | 56
Diarrhoea (Gastrointestinal disorders) | 49 | 9
Constipation (Gastrointestinal disorders) | 2 | 19
Mouth ulceration (Gastrointestinal disorders) | 6 | 3
Stomatitis (Gastrointestinal disorders) | 6 | 0
Leukopenia (Blood and lymphatic system disorders) | 7 | 51
Neutropenia (Blood and lymphatic system disorders) | 5 | 53
Anaemia (Blood and lymphatic system disorders) | 8 | 44
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 18
Rash (Skin and subcutaneous tissue disorders) | 78 | 11
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 7
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 10
Dry skin (Skin and subcutaneous tissue disorders) | 10 | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 9 | 0
White blood cell count decreased (Investigations) | 3 | 16
Alanine aminotransferase increased (Investigations) | 13 | 2
Platelet count decreased (Investigations) | 1 | 14
Aspartate aminotransferase increased (Investigations) | 11 | 3
Neutrophil count decreased (Investigations) | 2 | 10
Blood bilirubin increased (Investigations) | 11 | 0
Haemoglobin decreased (Investigations) | 0 | 6
Decreased appetite (Metabolism and nutrition disorders) | 14 | 30
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 7
Fatigue (General disorders) | 6 | 20
Pyrexia (General disorders) | 8 | 13
Chest discomfort (General disorders) | 6 | 3
Dizziness (Nervous system disorders) | 7 | 14
Headache (Nervous system disorders) | 5 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 19 | 9
Paronychia (Infections and infestations) | 17 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 6
Insomnia (Psychiatric disorders) | 5 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.